CLINICAL TRIAL: NCT07276503
Title: Predictors for the Development of Perioperative Delirium in Adult Patients Undergoing Elective Cardiac Surgery
Brief Title: Verification of a New Predictive Delirium Score in Adults With Elective Cardiac Valve or Bypass Surgery With Perioperative Use of a Heart-lung Machine; a Monocentric Pilot Observational Study
Acronym: MO-FA2-(TB)
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Verify-MO-FA2-(TB)
Record Dates: First submitted 2025-11-28; First posted 2025-12-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Emergence Delirium; Postoperative Delirium
Keywords: predicitve; delirium; postoperative; valve surgery; bypass surgery; Score; MO-FA2-(TB)
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adults with elective valve or bypass surgery using heart-lung machine

SUMMARY:
Basics (state of scientific knowledge):

Delirium is an acute disturbance of consciousness and attention that develops over a short period of time and fluctuates in severity. It is accompanied by a deterioration in cognitive performance, such as memory deficits, disorientation, and speech and thinking disorders, which significantly exceed the degree of any pre-existing limitations . Surgery and intensive medical treatment are considered to be two of the triggers.

In cardiac surgery, the incidence is reported to be between 10 and 50%, depending on the patient population. Delirium occurs approximately 3-4 days after surgery and lasts for several days. Relevant factors in the cardiac surgery population include age, duration of aortic clamping time or surgical technique, pre-existing conditions such as the extent of heart failure (EuroScore), diabetes mellitus, mental and cognitive impairments, or carotid stenosis.

Both current studies and current recommendations emphasize prevention and the lack of successful treatment options. Preventive measures are primarily investigated in packages of measures. The study presented here aims to define risk populations and test the sensitivity and specificity of the MO-FA2-(TB) score for the development of delirium.

Objectives of the study:

Verification of the predictive score "MO-FA2-(TB)" for the development of postoperative delirium Recording of delirium and associated influencing factors and endpoints

Categories examined in the score:

Memory using a list of words that must be memorized and repeated after a few minutes Orientation by asking about the year, month, date, day of the week, city, and location Frailty using the ASA score Use of heart-lung machine Incision-suture time

Study duration (for individual subjects):

postoperative intensive care stay up to and including day 10

Study population Patients who have to undergo cardiac surgery with CPB

Inclusion criteria:

Elective cardiac surgery Heart valve surgery, bypass surgery with CPB Length of stay in ICU > 48 hours Age ≥18 years Fluent German language skills

Exclusion criteria:

Age <18 years Lack of capacity to give consent Emergency Readmission to intensive care unit OPCAB surgery, microsurgical procedure

Recruitment: Information provided the day before surgery based on the surgical schedule If consent is given, score is recorded If ICU stay >48 hours, treatment data is recorded, otherwise exclusion Data collection up to and including d10

Treatment data collected:

Preoperative data, including ejection fraction, aids, abuse, scores collected ("4AT test" for rapid assessment of delirium and cognitive impairment, "MO-FA2-(TB)", "geriatric check" for identifying a geriatric patient) Intraoperative data, including duration of surgery, duration of heart-lung machine, acidosis Postoperative data in ICU, including delirium scores (ICDSC, CAM-ICU), days on ventilation, days of treatment, fluid intake, medication related to delirium, organ replacement therapy such as dialysis

Number of cases: Approx. 100 patients

Methodology Monocentric, observation

DETAILED DESCRIPTION:
The data listed below is collected from the PDMS if the patient has been in the ICU for more than 48 hours.

Master data and pre-existing conditions Age (at admission) Case number Gender Diagnosis Cardiac ejection fraction in % Type of surgery According to surgical protocol Dementia yes/no Hearing aid yes/no Glasses yes/no Abuse: nicotine, alcohol, drugs Premedication with benzodiazepines yes/no

Preoperative data 4AT test Collected yes/no, four factors MO-FA2-(TB) Detailed score Geriatric check Collected yes/no, result Deviation of surgical planning from surgical program Difference in surgical sites Planned duration of surgery Minutes

Intraoperative data pO2 Percentage drop below induction values Acidosis yes/no Number of pH < 7.3; Lactateemia: max lactate concentration nmol/l Maximum in mmol/l Actual surgery duration Minutes Duration of heart-lung machine Minutes Blood loss Number of blood units administered Type of anesthesia TIVA yes/no; conduction anesthesia (spinal, EDC, block)

Data collection in ICU Diagnosis of delirium (date) Recorded daily by ICDSC and CAM-ICU Delirium score >50%/d pos. / not recorded Daily Days/hours of ventilation Total in hours NIV >3x1.5h yes/no Days of treatment in ICU Total for > 2 days of stay in ICU Place of discharge (recorded on day 28) IMC/general ward (+sitting guard)/ext. Hospital/Rehab/Home ventilation/Death Fluid intake 24h Liters daily Organ replacement therapy Dialysis / Plasmapheresis daily Tracheotomy Yes/no / Days with tracheostoma Singer Index Number (discharge) Day with acidosis (50% <7.35) Daily Sofa score Daily Pregabalin, esketamine, oxycodone Daily NRS/VAS score or BPS/external assessment Score 3x/d >3 / 3x "shows pain"/manipulation Benzodiazepines Total requirement in ICU in mg Haloperidol, clonidine, quetiapine, etc. Per cumulative dose in mg/d Other: Risperidone, Clozapine, Pipamperone Per cumulative dose in mg/day Organ replacement procedures (dialysis, ECMO, ECLS, plasmapheresis) Number of days after organ replacement procedure Deceased on day 28/transferred Transfer/type of discharge

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery Heart valve surgery, bypass surgery with CPB
* Length of stay in ICU > 48 hours
* Age ≥18 years
* Fluent German language skills

Exclusion Criteria:

* Age <18 years
* Lack of capacity to give consent
* Emergency
* Readmission to intensive care unit
* OPCAB surgery, microsurgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with Elective cardiac surgery Heart valve surgery, bypass surgery with CPB
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-08 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients after heart surgery with postoperative delirium | from 48 hours ICU stay to day 10 of ICU stay or dismssal from ICU
  Relation between result of MO-FA2-(TB)-Score and actual development of postoperative delirium

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rosenberger, Prof. Dr., Study Director — Universitaetsklinikum Tuebingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez A, Thomas C, Deeken F, Wagner S, Kloppel S, Kentischer F, von Arnim CAF, Denkinger M, Conzelmann LO, Biermann-Stallwitz J, Joos S, Sturm H, Metz B, Auer R, Skrobik Y, Eschweiler GW, Rapp MA; PAWEL Study group. Patient safety, cost-effectiveness, and quality of life: reduction of delirium risk and postoperative cognitive dysfunction after elective procedures in older adults-study protocol for a stepped-wedge cluster randomized trial (PAWEL Study). Trials. 2019 Jan 21;20(1):71. doi: 10.1186/s13063-018-3148-8. PMID 30665435
- [Background] Wu SJ, Sharma N, Bauch A, Yang HC, Hect JL, Thomas C, Wagner S, Forstner BR, von Arnim CAF, Kaufmann T, Eschweiler GW, Wolfers T; PAWEL Study Group. Predicting Postoperative Delirium in Older Patients Before Elective Surgery: Multicenter Retrospective Cohort Study. JMIR Aging. 2025 Aug 19;8:e67958. doi: 10.2196/67958. PMID 40828691